CLINICAL TRIAL: NCT02253472
Title: The Safety and Efficacy of Long-term Treatment of PINS Stimulator System for Patients With Obsessive-Compulsive Disorder
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-008
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Stimulation is on.
  Interventions: Device: Deep Brain Stimulation
- Placebo (Sham Comparator): Stimulation is off.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation
  Other Names: Implanted device

SUMMARY:
The purpose of this clinical study is To verify the long term effectiveness and safety of a bilateral deep brain stimulation (DBS) produced by Beijing PINS Medical Co., Ltd. as a treatment option for patients with cognitive, behavioral, and functional disability of Obsessive-Compulsive Disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Obsessive compulsive disorder (according to DSM IV-criteria) as the primary psychiatric diagnosis.
2. Severity level of OCD more than 25 on the Yale-Brown Obsessive Compulsive Scale.
3. Course of illness had to have been present for at least five years in a chronic or progressive form despite any treatment trials (treatment resistance).
4. Treatment resistance: at least two serotonin reuptake inhibitors (SSRI´s), or one SSRI and clomipramine in 5.Sufficient dosages for at least 10 weeks, an augmentation trial with lithium, buspirone or a neuroleptic Lasting at least 10 weeks, and complete cognitive-behavioral psychotherapy, including "exposure and response Prevention" of a minimum of 20 sessions with a documented lack of efficiency.

6.The ability to give written and informed consent.

Exclusion Criteria:

1. Co-morbid psychotic disorder according to DSM-IV criteria
2. Suicidal tendencies in the last 6 months
3. History of cerebral trauma
4. Clinically relevant internal or neurological disorder
5. Substance misuse or dependence in the last six months
6. Ineligibility to fulfill the neurosurgical and anesthesiological preconditions for the implantation of a DBS
7. Participate in other clinical trial
8. The investigator and/or enrollment review committee, would preclude participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown obsessive-compulsive psychiatrists rating scale(Y-BOCS) | 12 month

SECONDARY OUTCOMES:
Hamilton anxiety scale (HAMD) | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University